CLINICAL TRIAL: NCT01591057
Title: Effect of Increased Fruit and Vegetable Intake on Biomarkers of Fruit and Vegetable Consumption
Brief Title: Effect of Fruit and Vegetable Intake on Markers of Fruit and Vegetable Consumption
Acronym: BIOFAV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Responsible Party: Principal Investigator, Jayne Woodside, PhD, Reader in Clinical Biochemistry, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 11/07
Record Dates: First submitted 2012-04-27; First posted 2012-05-03 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Healthy
Keywords: fruit; vegetables; biomarkers; randomised controlled feeding study; Fruit and vegetable intake biomarkers in healthy adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 2 Portions (Experimental)
  Interventions: Dietary Supplement: 2 portions of fruit and vegetables per day
- 5 portions (Experimental)
  Interventions: Dietary Supplement: 5 portions of fruit and vegetables per day
- 8 portions (Experimental)
  Interventions: Dietary Supplement: 8 portions of fruit and vegetables per day

INTERVENTIONS:
Dietary Supplement: 2 portions of fruit and vegetables per day — Consume 2 portions of fruit and vegetables per day
  Other Names: 2 portions/day
  Arms: 2 Portions
Dietary Supplement: 5 portions of fruit and vegetables per day — Consume 5 portions of fruit and vegetables per day
  Other Names: 5 portions/day
  Arms: 5 portions
Dietary Supplement: 8 portions of fruit and vegetables per day — Consume 8 portions of fruit and vegetables per day
  Other Names: 8 portions/day
  Arms: 8 portions

SUMMARY:
This study will examine what contribution of 'markers' of fruit and vegetable (FV) intake in blood and urine is most closely related to FV intake. 30 healthy volunteers will be fed either 2, 5 or 8 portions of FV per day for 4 weeks (ten participants per group, randomly assigned). Volunteers will have all their food provided during the study, and will consume two meals each weekday at the University. Volunteers will complete diet and lifestyle questionnaires at the start and end of the study and will have blood and urine samples collected at 0, 2 and 4 weeks.

DETAILED DESCRIPTION:
Single biomarkers of FV consumption, such as Vitamin C and certain carotenoids and flavonoids, have been proposed, but associations between these compounds and FV intake are relatively weak. The investigators propose that, given the complexity of FV, production of an algorithm based on a wide variety of bioactive compounds found in FV might better predict FV consumption. A controlled feeding study (30 volunteers randomised to 2, 5 or 8 portions of FV day for 4 weeks) will allow development of such an algorithm. Volunteers will be recruited by advertisement from QUB and the general public, and will have all their food provided for the 4 week period (two meals per day during the week to be consumed under supervision at the University).

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years
* Usual consumption of fruit and vegetables <= 2 portions/day

Exclusion Criteria:

* Use of any high dose vitamin, mineral or dietary supplements
* Current smoker
* BMI > 35 kg/m2
* Inability to provide informed consent
* Excessive alcohol consumption (>28 Units/week men or >21 Units/week women)
* Food sensitivities or allergies that would interfere with a tolerance of a fruit and vegetable rich diet
* Medical conditions or dietary restrictions that would substantially limit inability to complete the study requirements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Change in biomarkers of fruit and vegetable consumption | Baseline and 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jayne V Woodside, PhD, Principal Investigator — Queen's University, Belfast
Locations (1):
- Queen's University Belfast, Belfast, United Kingdom

REFERENCES:
- [Derived] Appleton KM, McGrath AJ, McKinley MC, Draffin CR, Hamill LL, Young IS, Woodside JV. The value of facial attractiveness for encouraging fruit and vegetable consumption: analyses from a randomized controlled trial. BMC Public Health. 2018 Mar 1;18(1):298. doi: 10.1186/s12889-018-5202-6. PMID 29490640
- [Derived] McGrath AJ, Hamill LL, Cardwell CR, Draffin CR, Neville CE, Appleton KM, McEneny J, McKinley MC, Young IS, Woodside JV. Combining vitamin C and carotenoid biomarkers better predicts fruit and vegetable intake than individual biomarkers in dietary intervention studies. Eur J Nutr. 2016 Jun;55(4):1377-88. doi: 10.1007/s00394-015-0953-7. Epub 2015 Jun 17. PMID 26081648